CLINICAL TRIAL: NCT05901623
Title: Neurodevelopmental Outcome of the Infants With Transient Hypothyroxinemia of Prematurity in Newborn Intensive Care Unit
Brief Title: ASQ Scores of Transient Hypothyroxinemia of Prematurity
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seda Yilmaz Semerci, Principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2022-20-05
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Transient Hypothyroxinemia of Prematurity; Neurodevelopmental Abnormality
MeSH Terms: interventions — Glycation End Products, Advanced; Equipment and Supplies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Infants with THoP
  Interventions: Other: 'Ages and Stages Questionnaries' (ASQ)
- Control: Healthy infants
  Interventions: Other: 'Ages and Stages Questionnaries' (ASQ)

INTERVENTIONS:
Other: 'Ages and Stages Questionnaries' (ASQ) — ''ASQ' is a screening tool for assessing the development of infants and preschoolers in the areas of communication, fine motor, gross motor, problem-solving and personal-social development, and 'ASQ:SE' is a screening tool for social-emotional development
  Other Names: 'Ages and Stages Questionnaries: Social-Emotional' (ASQ:SE) Inventories

SUMMARY:
• Transient hypothyroxinemia of prematurity (THoP) is defined as free thyroxine (FT4) level is below the reference values despite normal TSH level in preterm infant. This study aims to evaluate the neurological development of infants with transient premature hypothyroxinemia (THoP).

ELIGIBILITY:
Inclusion Criteria:

* newborn infants who were born at 28-36 gestational weeks
* Infants who were hospitalized in the neonatal intensive care unit
* Infants with transient hypothyroxinemia of prematurity

Exclusion Criteria:

* Newborns with maternal thyroid disease,
* Severe intracranial issues,
* Chromosomal and congenital anomalies,
* Infants older than 36 gestational weeks

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study included newborn infants born at 28-36 gestational weeks, with a diagnosis of transient hypothyroxinemia of prematurity, and hospitalized in the neonatal intensive care unit. Healthy age-matched infants were included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Long-term Neurodevelopment | 5 years
  'Ages And Stages Questionnaires' (ASQ) 'Ages And Stages Questionnaires: Social-Emotional' (ASQ:SE) Developmental Screening Tests evaluates the areas of communication, fine motor, gross motor, problem-solving and personal-social development. ASQ score differs 0-60 and results are interpreted in three group according to the gained points as normal, risky, and follow-up required.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No